CLINICAL TRIAL: NCT04938427
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Soticlestat as Adjunctive Therapy in Pediatric and Adult Subjects With Lennox-Gastaut Syndrome (LGS)
Brief Title: A Study of Soticlestat as an Add-on Therapy in Children, Teenagers, and Adults With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935-3002; 2021-002481-40 (EudraCT Number); jRCT2051210073 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-06-18; First posted 2021-06-24 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Lennox Gastaut Syndrome (LGS)
Keywords: Drug therapy
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — soticlestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Soticlestat placebo-matching mini-tablets or tablets, orally or via G-tube or MIC-KEY button or J-tube, BID, up to 4 weeks during titration. Participants continued to receive soticlestat placebo-matching mini-tablets or tablets for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period). Soticlestat matching tapering was done to maintain the blind if participants decided to discontinue the treatment.
  Interventions: Drug: Placebo
- Soticlestat (Experimental): Participants weighing <45 kg: Soticlestat, mini-tablets, at the dose of 40 mg to 200 mg, orally or via G-tube or MIC-KEY button or J-tube, BID based on body weight up to 4 weeks during titration. Participants continued to receive the dose that they were on at the end of the titration, for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period) with the dose tapered down if participants decided to discontinue the treatment.
  Participants weighing ≥45 kg: Soticlestat mini-tablets or tablets with a starting dose of 100 mg BID followed by 200 mg BID and, then 300 mg BID, up to 4 weeks during titration. Participants continued to receive 300 mg BID for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period) with the dose tapered down if participants decided to discontinue the treatment.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Placebo — Soticlestat placebo-matching mini-tablets or tablets.
  Arms: Placebo
Drug: Soticlestat — Soticlestat mini-tablets or tablets.
  Other Names: TAK-935
  Arms: Soticlestat

SUMMARY:
The aims of the study are:

* to learn if soticlestat, when given as add-on therapy, reduces the number of major motor drop seizures in children, teenagers, and adults with Lennox-Gastaut Syndrome.
* to assess the safety profile of soticlestat when given in combination with other therapies.

Participants will receive their standard antiseizure therapy, plus either tablets of soticlestat or placebo. A placebo looks just like soticlestat but will not have any medicine in it. Participants will take soticlestat or placebo for 16 weeks, followed by a gradual dose reduction for 1 week. Then, participants will be followed up for 2 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). Soticlestat will be assessed for efficacy, safety, and tolerability in pediatric and adult participants with LGS.

The study will enroll approximately 234 patients. Participants will be randomly assigned (by chance, like flipping a coin) in a 1:1 ratio to receive standard of care (SOC) plus one of the following adjunctive therapies which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

1. Soticlestat
2. Placebo (dummy inactive pill - this is a tablet/mini-tablet that looks like the study drug but has no active ingredient)

Participants will receive soticlestat or matching placebo based on their weight in the 4-week Titration Period. Following the Titration Period, participants will continue to receive the same dose in the 12-week Maintenance Period. The dose will then be down-tapered if participants decide to discontinue the treatment and/or are not deemed eligible to continue in Open-label extension (OLE).

This multi-center trial will be conducted worldwide. The overall time to participate in the study will be from 22-25 weeks. At the end of the treatment period, participants have the option to either complete the study and taper off the investigational product or to enter the OLE if they meet eligibility requirements. If participants discontinue, they will be followed-up on phone call approximately 14 days after the last dose of study drug for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Has documented clinical diagnosis of LGS.
2. Has had ≥8 MMD seizures each month in the 3 months prior to Screening based on the historical information and has had ≥8 MMD seizures per 28 days during the 4 to 6 week prospective Baseline Period.
3. Weighs ≥10 kg at the Screening Visit (Visit 1).
4. Failure to control seizures despite appropriate trials of at least 1 ASM based on historical information, and is currently on an antiseizure therapy or other treatment options considered as standard of care (SOC).
5. Artisanal cannabidiols are allowed at a stable dose for at least 4 weeks before the screening visit (Visit 1); the dosing regimen and manufacturer should remain constant throughout the study. (Artisanal cannabidiols will not be counted as ASMs.)
6. Currently taking 0 to 3 ASMs at stable doses for at least 4 weeks before the Screening Visit (Visit 1); Fenfluramine and cannabidiol (Epidiolex) are allowed where available and counted as an ASM. ASM dosing regimen must remain constant throughout the study.

Exclusion Criteria:

1. Admitted to a medical facility and intubated for treatment of status epilepticus 2 or more times in the 3 months immediately before Screening (Visit 1). For the purpose of this exclusion criterion, status is defined as continuous seizure activity lasting longer than 5 minutes or repeated seizures without return to Baseline in between seizures.
2. Unstable, clinically significant neurologic (other than the disease being studied), psychiatric, cardiovascular, ophthalmologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, endocrine disease, malignancy including progressive tumors, or other abnormality that may impact the ability to participate in the study or that may potentially confound the study results. It is the responsibility of the investigator to assess the clinical significance; however, consultation with the medical monitor may be warranted.
3. Considered by the investigator to be at imminent risk of suicide or injury to self, others, or property, or the participant has attempted suicide within 12 months before the Screening Visit (Visit 1). Participants who have positive answers on item numbers 4 or 5 on the Columbia suicide severity rating scale (C-SSRS) before dosing (Visit 2) are excluded. This scale will only be administered to participants aged ≥6 years.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (98):
- United States (24):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Center For Neurosciences, Tucson, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado., Denver, Colorado
  - Pediatric Neurology PA, Winter Park, Florida
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics - (CRS), Iowa City, Iowa
  - Midatlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Minnesota Epilepsy Group PA, Roseville, Minnesota
  - Institute of Neurology and Neurosurgery at Saint Barnabas, LLC, Livingston, New Jersey
  - Premier Healthcare Inc., New York, New York
  - NYU Comprehensive Epilepsy Center, New York, New York
  - Northwell Health Physician Partners - Neurology at Lenox Hill, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - WellSpan Oncology Research, York, Pennsylvania
  - Medical University of South Carolina Children Hospital - PIN, Charleston, South Carolina
  - Cook Children's Medical Center - Jane and John Justin Neurosciences Center, Fort Worth, Texas
  - University of Utah - Primary Children's Hospital - PPDS, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research & Innovation (Tacoma), Tacoma, Washington
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Belgium (3):
  - UZ Antwerpen PIN, Edegem, Antwerpen
  - Centre Neurologique William Lennox, Ottignies-Louvain-la-Neuve, Brabant Wallon
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels
- Canada (3):
  - Alberta Childrens Hospital, Calgary, Alberta
  - Child and Family Research Institute, Vancouver, British Columbia
  - Hospital For Sick Children, Toronto, Ontario
- China (12):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Women And Children's Medical Center, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Wuhan Childrens hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
- France (5):
  - CHRU Dijon Hopital General, Dijon, Cote-d'Or
  - Hopital Roger Salengro, Lille, Nord
  - Hopitaux de La Timone, Marseille
  - Hopital Necker - Enfants Malades, Paris
  - Hopital Robert Debre, Paris
- Germany (4):
  - Schon Klinik Vogtareuth, Vogtareuth, Bavaria
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Krankenhaus Mara gGmbH - Epilepsiezentrum Bethel, Bielefeld, North Rhine-Westphalia
  - Kleinwachau Sachsisches Epilepsiezentrum Radeberg Gemeinnutzige Gmbh, Radeberg, Sachse
- Greece (3):
  - Attikon University General Hospital, Chaïdári, Attica
  - University General Hospital of Larissa, Larissa
  - Hippokration Hospital, Thessaloniki
- Hungary (4):
  - Pecsi Tudomanyegyetem, Pécs, Baranya
  - Szent Janos Korhaz es Eszak-Budai Egyesitett Korhazak, Budapest
  - Bethesda Gyermekkorhaz, Budapest
  - Orszagos Mentalis, Ideggyogyaszati es Idegsebeszeti Intezet, Budapest
- Italy (4):
  - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - ASST di Pavia - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
- Japan (11):
  - Aichi Medical University Hospital, Nagakute-Shi, Aiti
  - Fukuoka Children's Hospital, Fukuoka, Hukuoka
  - Kumamoto-Ezuko Medical Center for The Severely Disabled, Kumamoto, Kumamoto
  - National Hospital Organization Nagasaki Medical Center, Omura-Shi, Nagasaki
  - National Hospital Organization Nishi-Niigata Chuo National Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Yasuhara Childrens Clinic, Neyagawa, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-Shi, Osaka
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
- Childrens University Hospital, Riga, Latvia
- Netherlands (2):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Stichting Epilepsie Instellingen Nederland, Zwolle, Overijssel
- Poland (3):
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny im. H.Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
- UGMK-Zdorojie, LLC, Yekaterinburg, Russia
- Serbia (4):
  - Clinic for Neurology and Psychiatry for Children and Youth, Belgrade
  - Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade
  - University Clinical Center Nis, Niš
  - Children and Youth Health Care Institute of Vojvodina, Novi Sad
- Spain (5):
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Regional Universitario de Malaga Hospital General, Málaga
  - Centro de Neurologia Avanzada, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (5):
  - Municipal Institution Dnipropetrovsk Regional Children Clinical Hospital of DRC, Dnipro, Dnipropetrovsk Oblast
  - Communal Non-profit Enterprise City Childrens Clinical Hospital #6 of DCC, Dnipro, Dnipropetrovsk Oblast
  - Communal Non-commercial Enterprise Iv-Frank Regional Childrens Clinical Hosp of Iv-Frank RC, Ivano-Frankivsk
  - CNPE Clinical Hospital Psychiatry of the Executive Body of the Kyiv City Council KCSA, Kyiv
  - SI Ukr. Med. Rehabilitation Center For Children With Organic Injury of Nervous System of MoH of Ukr, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/60e30ebd1f1122001e30a940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 84 investigative sites in Australia, Belgium, Canada, China, France, Germany, Greece, Hungary, Italy, Japan, Latvia, Netherlands, Poland, Russian Federation, Serbia, Spain, Ukraine and the United States from 08 November 2021 to 25 January 2024.
Pre-assignment Details: A total of 270 participants with a diagnosis of Lennox-Gastaut syndrome were randomized in a 1:1 ratio to receive either soticlestat or placebo.
Groups:
- Placebo: Soticlestat placebo-matching mini-tablets or tablets, orally or via gastrostomy tube (G-tube) or low-profile gastric tube (MIC-KEY) button or jejunostomy tube (J-tube), twice daily (BID), up to 4 weeks during titration. Participants continued to receive soticlestat placebo-matching mini-tablets or tablets for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period). Soticlestat matching tapering was done to maintain the blind if participants decided to discontinue the treatment.
- Soticlestat: Participants weighing <45 kilograms (kg): Soticlestat, mini-tablets, at the dose of 40 mg to 200 mg, orally or via G-tube or MIC-KEY button or J-tube, BID based on body weight up to 4 weeks during titration. Participants continued to receive the dose that they were on at the end of the titration, for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period) with the dose tapered down if participants decided to discontinue the treatment.
  Participants weighing ≥45 kg: Soticlestat mini-tablets or tablets with a starting dose of 100 mg BID followed by 200 mg BID and, then 300 mg BID, up to 4 weeks during titration. Participants continued to receive 300 mg BID for 12 weeks during maintenance. The total duration of the treatment was up to 16 weeks (Full Treatment Period) with the dose tapered down if participants decided to discontinue the treatment.
Period: Overall Study
Arm/Group | Placebo | Soticlestat
Started | 136 | 134
Completed | 126 | 114
Not Completed | 10 | 20
Not completed — Adverse Event | 5 | 19
Not completed — Withdrawal by Parent/Guardian | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Reason Not Specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Soticlestat | Total
Number analyzed (Participants) | 136 | 134 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (6.68) | 13.4 (9.35) | 12.9 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 52 | 55 | 107
  Gender: Male | 84 | 79 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 7 | 11
  Ethnicity: Not Hispanic or Latino | 130 | 124 | 254
  Ethnicity: Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 44 | 42 | 86
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: Black or African American | 2 | 1 | 3
  Race: White | 81 | 86 | 167
  Race: More than one race | 2 | 0 | 2
  Race: Unknown or Not Reported | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Major Motor Drop (MMD) Seizure Frequency Per 28 Days During the Full Treatment Period
Description: MMD seizure frequency per 28 days was defined as the total number of MMD seizures reported during the period divided by the number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the full Treatment Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Full Treatment Period: Weeks 1 to 16
Population: Modified Intent-to-treat (mITT) Analysis Set included all randomized participants who had received at least 1 dose of study drug and had been assessed for seizures for at least 1 day in the Full Treatment Period.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
percent change | -6.69 [-26.41 to 24.26] | -6.11 [-38.02 to 31.99]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.785, ANCOVA — The p-value was calculated using Rank Analysis of Covariance (ANCOVA) model using treatment group, age stratum (≤6 years, >6 years), and rank of Baseline seizure frequency per 28 days as predictors; Hodges-Lehmann Location Shift Estimate = -1.17, 95% CI 2-sided [-13.02 to 9.99] — The location shift between soticlestat and placebo (soticlestat - placebo) and its asymptotic 95% confidence interval (CI) are based on the Hodges-Lehmann estimation

2. Primary Outcome: Percent Change From Baseline in Major Motor Drop (MMD) Seizure Frequency Per 28 Days During the Maintenance Period
Description: MMD seizure frequency per 28 days was defined as the total number of MMD seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the Maintenance Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Maintenance Period: Weeks 5 to 16
Population: mITT Analysis Set included all randomized participants who had received at least 1 dose of study drug and had been assessed for seizures for at least 1 day in the Full Treatment Period. Overall number of participants analyzed indicates the number of participants with data available for analyses.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 132 | 124
percent change | -9.63 [-30.15 to 23.71] | -5.24 [-41.94 to 42.29]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; p = 0.778, ANCOVA — The p-value was calculated using the Rank ANCOVA model using the treatment group, age stratum (≤6 years, >6 years), and rank of Baseline seizure frequency per 28 days as predictors; Hodges-Lehmann Location Shift Estimate = 2.43, 95% CI 2-sided [-10.86 to 15.14] — The location shift between soticlestat and placebo (soticlestat - placebo) and its asymptotic 95% CI are based on the Hodges-Lehmann estimation

3. Secondary Outcome: Percentage of Responders During the Maintenance Period
Description: Responders are defined as those with ≥50% reduction from Baseline in MMD seizures during the Maintenance Period. Percentages are rounded off to the nearest single decimal place.
Time Frame: Maintenance Period: Weeks 5 to 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 132 | 124
percentage of participants | 11.4 | 19.4
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.94 to 3.87]

4. Secondary Outcome: Percentage of Responders During the Full Treatment Period
Description: Responders are defined as those with ≥50% reduction from Baseline in MMD seizures during the Full Treatment Period. Percentages are rounded off to the nearest single decimal place.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: mITT Analysis Set included all randomized participants who had received at least 1 dose of study drug and had been assessed for seizures for at least 1 day in the Full Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
percentage of participants | 9.6 | 16.4
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.92 to 4.05]

5. Secondary Outcome: Percentage of Participants With ≤0%, >0% to ≤25%, >25% to ≤50%, >50% to ≤75%, >75% to ≤100% Reduction in MMD Seizure During the Full Treatment Period
Description: Percent reduction from Baseline (%) is defined as [(Full Treatment Period MMD Seizure Frequency - Baseline MMD Seizure Frequency) divided by Baseline MMD Seizure Frequency] multiplied by 100. Data is reported as reduction of ≤0%, >0% to ≤25%, >25% to ≤50%, >50% to ≤75%, >75% to ≤100% or more in seizures from Baseline. Percentages are rounded off to the nearest single decimal place.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
percentage of participants
  ≤0% Reduction | 43.4 | 43.3
  >0% to ≤ 25% Reduction | 29.4 | 24.6
  >25% to ≤ 50% Reduction | 17.6 | 15.7
  >50% to ≤ 75% Reduction | 6.6 | 11.2
  >75% to ≤ 100% Reduction | 2.9 | 5.2

6. Secondary Outcome: Percentage of Participants With Caregiver Global Impression of Improvement (Care GI-I) Scale Responses as Per the Parent/Caregiver Reported Impression at Week 16
Description: The Care GI-I is a 7-point Likert scale that the caregiver used to rate improvement in overall seizure control, behavior, safety and tolerability after the initiation of study drug relative to Baseline (before treatment with the study drug). The participant was rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). The parent/caregiver completed the Care GI-I via interview. Lower scores indicate improvement. Percentages are rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 130 | 122
percentage of participants
  Score 1: Very Much Improved | 0.8 | 1.6
  Score 2: Much Improved | 13.1 | 20.5
  Score 3: Minimally Improved | 25.4 | 26.2
  Score 4: No Change | 46.2 | 36.9
  Score 5: Minimally Worse | 11.5 | 6.6
  Score 6: Much Worse | 3.1 | 5.7
  Score 7: Very Much Worse | 0.0 | 2.5
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.86 to 2.13]

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression of Improvement (CGI-I) Scale Responses as Per the Investigator Reported Impression at Week 16
Description: The CGI-I (Clinician) is a 7-point Likert scale that the investigator to rate a participant's change (improvement) in overall seizure control, behavior, safety and tolerability after the initiation of study drug relative to Baseline (before treatment with the study drug). The participant was rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). The investigator or designee will complete the CGI-I. Lower scores indicate improvement. Percentages are rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 133 | 132
percentage of participants
  Score 1: Very Much Improved | 1.5 | 3.0
  Score 2: Much Improved | 11.3 | 15.9
  Score 3: Minimally Improved | 17.3 | 24.2
  Score 4: No Change | 60.2 | 43.2
  Score 5: Minimally Worse | 5.3 | 7.6
  Score 6: Much Worse | 4.5 | 4.5
  Score 7: Very Much Worse | 0.0 | 1.5
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.89 to 2.21]

8. Secondary Outcome: Percentage of Participants With CGI-I Nonseizure Symptoms Instrument Responses for Each Domain as Per the Investigator Reported Impression at Week 16
Description: The CGI-I nonseizure symptoms instrument is a series of single-item assessments that the investigator used to rate improvement in the symptoms and impacts in select nonseizure domains (alertness, communication, and disruptive behaviors) since initiating the study drug. The participant was rated by the investigator for each domain as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). Lower scores indicated improvement. Data for percentage of participants categorized based on the responses for each domain are presented. Percentages are rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 133 | 132
percentage of participants
  Alertness: Score 1: Very Much Improved | 1.5 | 1.5
  Alertness: Score 2: Much Improved | 7.5 | 13.6
  Alertness: Score 3: Minimally Improved | 12.8 | 16.7
  Alertness: Score 4: No Change | 71.4 | 59.1
  Alertness: Score 5: Minimally Worse | 4.5 | 8.3
  Alertness: Score 6: Much Worse | 2.3 | 0.8
  Alertness: Score 7: Very Much Worse | 0.0 | 0.0
  Communication: Score 1: Very Much Improved | 1.5 | 2.3
  Communication: Score 2: Much Improved | 7.5 | 10.6
  Communication: Score 3: Minimally improved | 12.8 | 18.9
  Communication: Score 4: No Change | 71.4 | 61.4
  Communication: Score 5: Minimally Worse | 4.5 | 6.1
  Communication: Score 6: Much Worse | 2.3 | 0.8
  Communication: Score 7: Very Much Worse | 0.0 | 0.0
  Disruptive Behaviors: Score 1: Very Much Improved | 0.0 | 1.5
  Disruptive Behaviors: Score 2: Much Improved | 1.5 | 6.1
  Disruptive Behaviors: Score 3: Minimally improved | 8.3 | 10.6
  Disruptive Behaviors: Score 4: No Change | 79.7 | 75.0
  Disruptive Behaviors: Score 5: Minimally Worse | 6.8 | 3.8
  Disruptive Behaviors: Score 6: Much Worse | 3.8 | 2.3
  Disruptive Behaviors: Score 7: Very Much Worse | 0.0 | 0.8
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Alertness Domain; Test type: Superiority; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.85 to 2.30]
Statistical Analysis 2: Comparison: Placebo vs Soticlestat; Communication Domain; Test type: Superiority; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.91 to 2.48]
Statistical Analysis 3: Comparison: Placebo vs Soticlestat; Disruptive Behaviors Domain; Test type: Superiority; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.06 to 3.43]

9. Secondary Outcome: Change From Baseline in Quality of Life Inventory-Disability (QI-Disability) Total Score at Week 16
Description: The QI-Disability tool is a parent/caregiver-reported questionnaire evaluated the quality of life in children with intellectual disabilities. It contains 32 items covering 6 domains of quality of life: physical health, positive emotions, negative emotions, social interaction, leisure and the outdoors, and independence. Each QI-Disability item is rated on a Likert scale of: Never, Rarely, Sometimes, Often, and Very Often. Items were linearly transformed to a scale of 0 to 100, with higher scores representing better quality of life. Domain scores are calculated by averaging item scores. The domain scores are summed and divided by 6 to yield a total score. The total score ranges from 0 to 100, with higher scores indicating a better quality of life. A negative change from Baseline implies deteriorating quality of life. Mixed-effects model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 112 | 107
score on a scale | -1.66 (10.314) | -1.17 (12.042)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Least Square Mean Difference = 0.52, 95% CI 2-sided [-2.20 to 3.24]

10. Secondary Outcome: Percentage of Participants With CGI-I Seizure Intensity and Duration Instrument Responses as Per the Parent/Caregiver Reported Impression at Week 16
Description: The CGI-I seizure intensity and duration instrument was used by the parent/caregiver to rate changes in intensity and/or duration of the most impactful seizures from the first assessment. The participant's symptoms were rated as follows: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), and 7 (very much worse). Lower scores indicate improvement. Percentages are rounded off to the nearest single decimal place.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 131 | 122
percentage of participants
  Score 1: Very Much Improved | 0.8 | 1.6
  Score 2: Much Improved | 9.9 | 18.9
  Score 3: Minimally Improved | 24.4 | 28.7
  Score 4: No Change | 51.1 | 39.3
  Score 5: Minimally Worse | 9.9 | 4.1
  Score 6: Much Worse | 3.8 | 5.7
  Score 7: Very Much Worse | 0.0 | 1.6
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.06 to 2.65]

11. Secondary Outcome: Percent Change From Baseline in Frequency of All Seizures Per 28 Days During the Maintenance Period
Description: Seizure frequency per 28 days was defined as the total number of seizures reported during the period divided by the number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the Maintenance Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Maintenance Period: Weeks 5 to 16
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 132 | 124
percent change | -9.92 [-30.55 to 15.55] | -16.82 [-40.93 to 20.60]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Hodges-Lehmann Location Shift Estimate = -6.37, 95% CI 2-sided [-16.83 to 4.16] — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Percent Change From Baseline in Frequency of All Seizures Per 28 Days During the Full Treatment Period
Description: Seizure frequency per 28 days was defined as the total number of seizures reported during the period divided by the number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline was defined as (frequency of seizures per 28 days during the full Treatment Period - frequency of seizures per 28 days at Baseline) divided by the frequency of seizures per 28 days at Baseline multiplied by 100.
Time Frame: Baseline; Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
percent change | -6.45 [-28.11 to 16.16] | -16.71 [-39.84 to 18.53]
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; Hodges-Lehmann Location Shift Estimate = -6.65, 95% CI 2-sided [-16.67 to 3.12] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Change From Baseline in Percentage of MMD Seizure-free Days During the Full Treatment Period
Description: MMD Seizure-free days was defined as the number of days the participant remained MMD seizure free after initiation of the treatment. The change from baseline in percentage of MMD seizure-free days, was defined as the percentage of seizure-free days during the Full Treatment Period minus the percentage of seizure-free days during the Baseline. A linear model with treatment group and age stratum as factors and baseline percentage as a covariate was used for analysis.
Time Frame: Baseline up to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
percentage of days | 5.37 (1.661) | 7.84 (1.676)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; LS Mean Difference = 2.47, 95% CI 2-sided [-1.74 to 6.67] — A linear model with treatment group and age stratum as factors and baseline percentage as a covariate was used for analysis

14. Secondary Outcome: Longest MMD Seizure-free Interval During the Full Treatment Period
Description: Longest MMD Seizure-free Interval was defined as the longest time period that the participant remained MMD seizure-free after initiation of the treatment. A linear model with treatment group and age stratum as factors was used for analysis.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
days | 5.5 (1.39) | 10.9 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; LS Mean Difference = 5.4, 95% CI 2-sided [1.9 to 8.9]

15. Secondary Outcome: Number of Days When Rescue Antiseizure Medication (ASM) is Used During the Full Treatment Period
Description: Use of rescue ASM was recorded in the case report form (CRF) along with start and end date of medication. Based on
  the start and end dates for all rescue ASMs taken by a participant, the number of days during the Full Treatment Period when rescue ASM was used was derived.
Time Frame: Full Treatment Period: Weeks 1 to 16
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Soticlestat
Number analyzed (Participants) | 136 | 134
days | 3.4 (1.12) | 2.5 (1.14)
Statistical Analysis 1: Comparison: Placebo vs Soticlestat; Test type: Superiority; LS Mean Difference = -0.9, 95% CI 2-sided [-3.7 to 2.0]

ADVERSE EVENTS:
Time Frame: From the first dose up to Week 19
Description: Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Arm/Group | Placebo | Soticlestat
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/134
Serious Adverse Events (participants affected / at risk) | 10/136 | 11/134
Other Adverse Events (participants affected / at risk) | 51/136 | 69/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=136) | Soticlestat (N=134)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Change in seizure presentation (Nervous system disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Negative pressure pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 2
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=136) | Soticlestat (N=134)
COVID-19 (Infections and infestations) | 3 | 8
Change in seizure presentation (Nervous system disorders) | 7 | 17
Constipation (Gastrointestinal disorders) | 3 | 7
Decreased appetite (Metabolism and nutrition disorders) | 3 | 8
Fall (Injury, poisoning and procedural complications) | 5 | 7
Fatigue (General disorders) | 5 | 8
Nasopharyngitis (Infections and infestations) | 11 | 10
Pyrexia (General disorders) | 11 | 10
Somnolence (Nervous system disorders) | 10 | 19
Upper respiratory tract infection (Infections and infestations) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT04938427/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT04938427/SAP_001.pdf